CLINICAL TRIAL: NCT01687530
Title: Randomised Controlled Trial to Evaluate the Safety Performance and Initial Efficacy of a Guided Bone Regeneration Membrane for the Treatment of Proximal (Subtrochanteric) Femoral Fractures
Brief Title: Evaluation of the Safety and Efficacy of a Guided Bone Regeneration Membrane for the Treatment of Femoral Fractures
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RegeneCure, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGO01/12
Record Dates: First submitted 2012-09-09; First posted 2012-09-19 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Proximal (Subtrochanteric)Femoral Fractures; Distal Femoral Fractures
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMCA bone membrane (Experimental): AMCA Bone is manufactured from Polyethylene Glycol 400 and Ammonio Methacrylate copolymer type A (Eudragit RL 100) materials.
  Interventions: Procedure: AMCA Bone Membrane.

INTERVENTIONS:
Procedure: AMCA Bone Membrane. — AMCA Bone Membrane, as a bone stimulating aid for orthopedic trauma applications.

SUMMARY:
Certain types of fractures require surgical intervention that may involve the use of bone grafts or bone graft substitutes. Many of the materials used as bone graft substitutes suffer from disadvantages such as soft tissue invasion of the fracture area, inadequate blood supply, failure to encourage the production of bone and ectopic bone formation.

A guided bone regeneration (GBR) environment may help in solving these clinical concerns. GBR has been widely used in the field of dentistry since the 1980s to provide stable placement for dental implants

The purpose of this study is to evaluate the safety, performance and initial efficacy of Regenecure's, AMCA Bone Membrane, as a bone stimulating aid for orthopedic trauma applications.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years
2. Both males and females
3. Females of child-bearing potential who have a negative urine hCG pregnancy test following informed consent and prior to surgical procedure and who are not planning to become pregnant for the duration of their part in the study
4. Femoral subtrochanteric fracture. The fracture is classified as one of the following:

   A. Closed fracture B. AO 31 A3, 33b + C1 + C2, and extending to the distal third
5. Proximal subtrochanteric femoral fracture will be treated with a cephalomedullary nail.
6. Patients must be available for follow-up for a minimum of 12 months.

Exclusion Criteria:

1. Trauma presentation

   * Open fractures
   * Bilateral fractures
   * Polytrauma with head injury
   * Presence of periprosthetic fractures
2. Patient Medical History

   * Previous malignancy (except basal cell carcinoma of the skin)
   * Active autoimmune disease
   * Metabolic bone disease (primary or secondary)
   * Chronic renal insufficiency (defined by a Glomerular Filtration Rate of <30 ml/min)
   * Liver function abnormality (defined by presence of ALT or AST levels more than double the upper limit)
   * Current smoker
3. Concurrent medication

   o Medications that may interfere with bone metabolism including:
4. Calcitonin for 7 days or more within the last 6 months prior to study
5. Bisphosphonates for 30 days or more within the last 12 months prior to study
6. Bone therapeutic doses of vitamin D or vitamin D metabolites for 30 days or more within the last 6 months

   * Previous or present immunosuppressive treatment
   * Previous radiotherapy or chemotherapy
   * Cumulative dose of 150mg total prednisolone or any other gluco-corticosteroid for 7 days or more within the last 6 months prior to study
   * Previous history of or current alcohol abuse
   * Previous history of or current drug addiction/abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the safety of the AMCA Bone membrane when used in the treatment of subtrochanteric femoral fractures. | 12 months
  Safety element will be measured by evaluation of swelling, clinical signs of superficial or deep infection, pain in the operated area.
  Radiographic healing assessment score.

SECONDARY OUTCOMES:
To evaluate the performance of the AMCA Bone membrane in providing enhanced healing of compromised fractures at risk of non-union. | 12 months
  efficacy will be assessed by radiographic evaluation and functional assessment at different time points.
  To evaluate the performance of the AMCA Bone membrane in providing enhanced healing of compromised fractures at risk of non-union, assessed by a difference of ten points in reduction of the completed Harris hip score at 16 weeks from baseline.

OTHER OUTCOMES:
To evaluate the performance of the AMCA Bone membrane in providing enhanced healing of compromised fractures at risk of non-union, assessed by a User Satisfaction | 12 months
  User Satisfaction, Usability Lack of side effects Reduction of the incidences rate of secondary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Amal Khoury, M.D, Study Director — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Hadassah Medical Organization, Orthopedic Surgery Department, Jerusalem
  - Orthopedic Department, Hadassah Medical Organization, Jerusalem